CLINICAL TRIAL: NCT02594267
Title: A Phase 1, Dose-Finding Study of Folotyn® (Pralatrexate Injection) Plus Cyclophosphamide, Doxorubicin, Vincristine, and Prednisone (CHOP) in Patients With Peripheral T-Cell Lymphoma (PTCL)
Brief Title: A Dose-Finding Study of Folotyn® (Pralatrexate Injection) Plus CHOP With Peripheral T-Cell Lymphoma (PTCL)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Acrotech Biopharma Inc. (Industry)
Collaborators: Axis Clinicals Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPI-FOL-101
Record Dates: First submitted 2015-09-25; First posted 2015-11-03 (Estimated); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Peripheral T-Cell Lymphoma (PTCL)
Keywords: PTCL; Peripheral T-Cell Lymphoma; Folotyn; Pralatrexate; CHOP
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — 10-propargyl-10-deazaaminopterin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Part 1: Dose Finding, Cohort 1 (Experimental): Dose finding Phase Intervention: Folotyn (Pralatrexate Injection) CHOP: Cyclophosphamide, Doxorubicin, Vincristine, and Prednisone
  The first cohort will begin with three patients with dose A of pralatrexate plus CHOP at full dose.
  The second cohort will begin with three patients with dose B of pralatrexate plus CHOP at full dose.
  The third cohort will begin with three patients with dose C of pralatrexate plus CHOP at full dose.
  The fourth cohort will begin with three patients with dose D of pralatrexate plus CHOP at full dose.
  The fifth cohort will begin with three patients with dose E of pralatrexate plus CHOP at full dose.
  Part 2: Dose Expansion, Additional ten patients will be enrolled at the MTD or MAD (if the MTD is not reached) plus CHOP at full dose in this part of the study. Blood samples for PK analysis of pralatrexate will be collected at various intervals pre and post pralatrexate injection during cycle 1, Dose 1.
  Interventions: Drug: Pralatrexate Injection

INTERVENTIONS:
Drug: Pralatrexate Injection — Drug: Folotyn (Pralatrexate Injection)
  CHOP : Cyclophosphamide, Doxorubicin, Vincristine, & Prednisone
  Other Names: Folotyn

SUMMARY:
The purpose of this study is to evaluate the Maximum Tolerated Dose (MTD) of pralatrexate in combination with cyclophosphamide, doxorubicin, vincristine, and prednisone (CHOP) regimen in patients with newly diagnosed peripheral T-cell lymphoma (PTCL).

DETAILED DESCRIPTION:
This is a Phase 1, open-label, multicenter, two-part, dose-finding, dose-escalation study.

The study is divided into two parts:

Part 1

Up to five sequential dose cohorts will enroll a maximum of 6 patients each. Escalation of the pralatrexate dose, after CHOP administration (Fol-CHOP), will continue in a traditional 3+3 design, until determination of the MTD. If the MTD is not reached, the Maximum Administered Dose (MAD) of pralatrexate in combination with CHOP will be 30 mg/m2 IV on Days 1 and 8 of each 21-day cycle for up to 6 cycles.

The first cohort will begin with three patients with dose A and CHOP at full dose. If none of the first three patients experiences a Dose-Limiting Toxicity (DLT), the next three patients will be enrolled in next higher dose cohort. If one of the first three patients in the first cohort experiences DLTs, an additional three patients will be enrolled into that cohort. If 2 or 3 of the first 3 patients experience DLTs, then the MTD is not found.

For cohorts 2, 3, 4, and 5, If none of the first three patients experiences a DLT, the next three patients will be enrolled in next higher dose cohort. If one of the first three patients in the first cohort experiences DLTs, an additional three patients will be enrolled into that cohort. If 2 or 3 of the first 3 patients experience DLTs, then the previous cohort will be considered the MTD and up to an additional 10 patients will be enrolled at that dose in Part 2 of the study.

Part 2

Once the MTD for the Fol-CHOP regimen has been established in Part 1 of the study, an additional 10 patients will be treated at the MTD (or MAD if MTD not reached) to confirm tolerability. Additionally, the PK of the established MTD of pralatrexate, when administered with CHOP at full dose, will be evaluated in these 10 patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or above
2. Adequate hematologic, hepatic, and renal function
3. Histologically confirmed, new diagnosis of PTCL
4. Eligible for CHOP regimen
5. Measurable disease based on Cheson 2007 criteria
6. Eastern Cooperative Oncology Group (ECOG) performance status < 2
7. Willing to perform at least two methods of contraception
8. Negative pregnancy test of females with childbearing potential.

Exclusion Criteria:

1. Active concurrent malignancy (except non melanoma skin cancer or carcinoma in situ of the cervix) or life threatening disease. If there is a history of prior malignancies or life threatening diseases, the patient must be disease free for at least 5 years.
2. Congestive heart failure Class III/IV according to the New York Heart Association (NYHA) Functional Classification.
3. Uncontrolled hypertension
4. Central nervous system (CNS) metastases .
5. Active uncontrolled infection, underlying medical condition, or other serious illness that would impair the ability of the patient to receive protocol treatment
6. Major surgery within 30 days prior to enrollment.
7. Use of any investigational drugs, biologics, or devices within 30 days prior or during the study treatment.
8. Previous exposure to pralatrexate.
9. Pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2015-11-10 (Actual); Primary Completion 2017-04-07 (Actual); Study Completion 2020-10-08 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | 126 Days
  To evaluate the Maximum Tolerated Dose (MTD) of pralatrexate in combination with cyclophosphamide, doxorubicin, vincristine, and prednisone (CHOP) regimen in patients with newly diagnosed peripheral T-cell lymphoma (PTCL)

SECONDARY OUTCOMES:
Number of participants with treatment emergent adverse events (TEAEs) using CTCAE version 4.03 | 126 Days
  Investigator will question the patient at every visit about AEs and intercurrent illnesses.
Objective Response Rate | 126 Days
  To evaluate the Objective Response Rate (ORR) of 6 cycles of Fol-CHOP
Plasma concentration of pralatrexate in combination with CHOP | 126 Days
  Measure the concentration of pralatrexate to evaluate the pharmacokinetics of pralatrexate when given in combination with CHOP using non-compartmental analysis.
Pharmacokinetics: Area Under the Curve (AUC) | 126 Days
  Non-compartmental Analysis
Pharmacokinetics: Maximum Concentration (Cmax) | 126 Days
  Non-compartmental Analysis
Pharmacokinetics: Time to Maximum concentration (Tmax) | 126 Days
  Non-compartmental Analysis
Pharmacokinetics: Clearance (CL) | 126 Days
  Non-compartmental Analysis

CONTACTS AND LOCATIONS:
Overall Officials: Erard Gilles, MD, Study Director — Navitas Life Sciences Inc.
Locations (4):
- United States (4):
  - Mayo Clinic, Rochester, Minnesota
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - MD Anderson, Houston, Texas
  - Seattle Cancer Care Alliance/University of Washington, Seattle, Washington

REFERENCES:
- [Derived] Iyer SP, Johnston PB, Barta SK. Pralatrexate injection combined with CHOP for treatment of PTCL: results from the Fol-CHOP dose-finding phase 1 trial. Blood Adv. 2024 Jan 23;8(2):353-364. doi: 10.1182/bloodadvances.2023011095. PMID 38029357